CLINICAL TRIAL: NCT07004582
Title: Preclinical ex Vivo Patient-derived 3D Cultures for the Prediction of Prostate Cancer Treatment Response
Brief Title: Lab Research Using Mini-tumors to Study Prostate Cancer Treatments
Acronym: PR3DICT
Status: Not yet recruiting | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Zuyderland Medical Centre (Other); Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: PR3DICT; NL-009852 (Registry Identifier: CCMO)
Record Dates: First submitted 2025-05-15; First posted 2025-06-04 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer; Prostate Cancer Metastatic Disease; Prostate Cancer Recurrent; Advanced Prostate Cancer
Keywords: Advanced prostate cancer; Metastatic prostate cancer; Prostate cancer; Patient-tailored treatment; Precision Medicine; Ex vivo prediction platform; Personalized medicine; Drug Screening Assays; Three-Dimensional Culture Techniques; Organoids; Tumoroids; Tumor replicas; Prostatic Neoplasms; Neoplasm Metastasis; Advanced Cancer; Treatment Outcome; Human Tissue Culture Techniques
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Prostate cancer tissue and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HDR brachytherapy: High-risk or recurrent prostate cancer patients that will undergo high dose rate (HDR) brachytherapy.
  Interventions: Procedure: HDR brachytherapy
- Diagnostic biopsy: Patients with MRI-suspected metastatic prostate cancer - with at least clinical stage T3-4 disease - that will undergo a diagnostic transperineal prostate biopsy procedure guided with ultrasound (i.e., targeted or template prostate cancer needle biopsies taken through the perineum guided with transrectal ultrasound)
  Interventions: Diagnostic Test: Diagnostic biopsy

INTERVENTIONS:
Procedure: HDR brachytherapy — High dose rate (HDR) brachytherapy for the treatment of high-risk or recurrent prostate cancer
  Groups: HDR brachytherapy
Diagnostic Test: Diagnostic biopsy — Transperineal prostate biopsies guided with transrectal ultrasound for the diagnosis of (recurrent) prostate cancer
  Groups: Diagnostic biopsy

SUMMARY:
For men with an aggressive form of prostate cancer, finding the right and effective treatment right away is challenging. Many of these men face a high risk of cancer recurrence: about half experience a relapse after surgery, and more than a third after undergoing radiation therapy. Men with metastatic prostate cancer have particularly poor prognoses, with a five-year survival rate of only 30% to 50%. In short, it is difficult to predict which treatment, or combination of treatments, will lead to longer survival for this group of men with aggressive (metastatic) prostate cancer.

In the laboratory, it is possible to grow small samples of tumors into 3D mini-tumors. These mini-tumors retain the characteristics of the patient's original tumor tissue. Various treatments can be tested on these 3D mini-tumors to determine which therapy is most effective for each individual case. There are currently two techniques available for creating these 3D mini-tumors in the lab. In this project, we aim to investigate which of these two techniques works best in order to test and personalize treatments.

DETAILED DESCRIPTION:
The biological diversity of high-risk prostate cancer makes it difficult to find an effective first-line or second-line cancer treatment. Therapy failure is high for men with high-risk localized cancer, having a risk of a biochemical relapse between 42% and 50% following radical prostatectomy and 36-43% after radiation therapy. Moreover, very high-risk prostate cancers with distant metastasis, accounting for 22% of the prostate cancer diagnoses, have a worse prognosis with overall 5-year survival rates of only 30-45%. Personalized treatment plans based on ex vivo therapy testing on patient-derived prostate cancer cultures could offer a more tailored approach by predicting the most effective therapy for each patient's specific tumor profile.

Ex vivo patient-derived 3D cultures may be an excellent solution which is able to recapitulate histological characteristics of the original tumor and could be utilized to assess tumorigenesis, potential drug targets and patients' drug responsiveness. Aside from the preservation of histological characteristics of the original tumor, ex vivo patient-derived 3D cultures are able to maintain physiological tumor features by preservation of the tumor micro-environment which is essential for testing selected types of anti-cancer drugs. Ex vivo patient-derived 3D cultures are generated from small fragments of tumor tissue containing organ-specific (tumor) cell types, which are cultivated into miniature, self-organizing prostate tumors using one of two principal techniques: organoid (i.e., utilizing a basement membrane exact) or tumor replica technology (i.e., utilizing a suspension culture without matrix support). Success rates of culturing prostate cancer organoids based on left-over tissue after radical prostatectomy are excellent, varying between 90% and 98%, however, for the more high-risk (metastasized) prostate cancers, the success rates vary considerably from 16% to 44% based on the small amount of needle biopsy tissue and inherent low cellular yield, limited cell-cell interaction, or prostate cancer subtype specific growth factors.

To overcome the above-mentioned low success-rates, the high turnaround time, and challenges of deriving (metastasized) prostate cancer organoids, the tumor replica technology may be interesting to explore. The tumor replica technology is optimized by Rianne Vaes at the Maastro Lab in the IPON-3 study for lung cancer (NL79010.068.21) and has increased the success rate from 17% to 70% (unpublished). So far, only one study generated prostate cancer tumor replicas utilizing this technique and showed an excellent success rate of 100% after radical prostatectomy. However, the establishment and use of tumor replicas derived from high-risk (metastatic) prostate cancer biopsies have been described yet, nor have been from prostate cancer recurrence following initial radiation therapy (i.e. radioresistant prostate cancer). Moreover, only one study demonstrated the capability of predicting the therapy response for prostate cancer drugs as well as radiation therapy on patient-derived 3D organoids of treatment-naïve prostate cancer patients utilizing left-over prostatectomy tissue. The number of patients on which treatment responsiveness was tested, however, was low (3 patients tested for prostate cancer drugs and 2 for radiation therapy).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Patients with prostate cancer
* Patients planned for HDR brachytherapy treatment for high-risk or recurrent prostate cancer or transperineal prostate biopsy with MRI-suspected metastatic prostate cancer with at least clinical stage T3-4.

Exclusion Criteria:

* Patients younger than 18 years
* Patients of whom it is not possible to obtain left-over tissue as part of the normal clinical treatment procedure (e.g., if all tumor material is required for the pathologist to make a diagnosis, to stage the patient or to perform a molecular diagnosis).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients planned for HDR brachytherapy treatment for high-risk or recurrent prostate cancer or transperineal prostate biopsy with MRI-suspected metastatic prostate cancer with at least clinical stage T3-4.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2031-09-30 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
Success rate | 1 year
  Determine the success rate of the established ex vivo prostate cancer 3D cultures from patient-derived (tumor) tissue material in which at least one first-line or second-line prostate cancer treatment (encompassing radiation exposure or cancer drugs) has been tested for sensitivity within a clinically relevant timeframe (up to 2 months).

SECONDARY OUTCOMES:
Most successful culturing technique per subtype | 1 year
  Evaluate the most successful culturing technique (organoid versus tumor replica) per prostate cancer subtype (e.g., different morphologies such as adenocarcinoma, carcinoid or neuroendocrine features; various tumor stages) for generating ex vivo patient-derived prostate cancer 3D cultures from biopsy tissue along with subsequent testing of first-line, second-line or novel/personalized prostate cancer treatments.
(epi)genetic and phenotypic tumor features | 1 year
  To investigate the stability of (epi-) genetic and phenotypic tumor features of patient-derived 3D prostate cancer cultures compared to the tumor of origin using, for example, H&E staining or immunohistochemistry stainings.
Treatment response | 5 years
  Compare the preclinical ex vivo patient-derived prostate cancer 3D culture predicted treatment sensitivity to prostate cancer drugs and/or radiation therapy to the patient clinical response, if possible.

CONTACTS AND LOCATIONS:
Overall Officials: Evert J Van Limbergen, PhD, MD, Principal Investigator — Maastricht Radiation Oncology
Locations (3):
- Netherlands (3):
  - Zuyderland Medisch Centrum, Heerlen, Limburg
  - Academisch Ziekenhuis Maastricht, Maastricht, Limburg
  - Maastricht Radiation Oncology, Maastricht, Limburg

IPD SHARING:
Plan to Share IPD: No
To protect participant privacy, individual patient-level data will not be shared. However, anonymized and de-identified data may be made available upon reasonable request, in accordance with applicable data protection regulations and institutional policies.